CLINICAL TRIAL: NCT01491490
Title: A Randomised, Doubleblind,Placebo Controlled, Parallel Group, Pilot Study of 40:1 Ratio of Formulated GW42003 :GW42004 in the Treatment of Iatrogenic Weight Gain and Dyslipidaemia Associated With Olanzapine Treatment in Subjects With Functional Psychosis
Brief Title: Treatment on Iatrogenic Weight Gain and Dyslipidaemia Associated With Olanzapine
Acronym: GWMD09126
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Chief Investigator and the Sponsor have concluded that it will not be possible to complete the enrolment in any meaningful timeframe.
Sponsor: GW Research Ltd (Industry)
Responsible Party: Sponsor
Organization: GWResearch (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWMD09126
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Functional psychosis; Schizophreniform; Acute psychosis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GWP42003 : GWP42004 (40:1) (Active Comparator)
  Interventions: Drug: GWP42003 : GWP42004 (40:1)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003 : GWP42004 (40:1) — Capsules taken once a day for 6 weeks
  Arms: GWP42003 : GWP42004 (40:1)
Drug: Placebo — Capsules taken once a day for 6 weeks
  Arms: Placebo

SUMMARY:
Olanzapine is one of the most effective and best tolerated of the atypical antipsychotics, but it is also particularly associated with weight gain and metabolic problems.

This study is being conducted by GW Pharma Ltd as a pilot study in order to determine the efficacy and safety of two medications GW42003 and GW42004 as a 40:1 ratio when combined with the subjects existing treatment of olanzapine in subjects with weight gain attributable to olanzapine treatment for functional psychosis. This is the first study to determine whether the study medications have a positive benefit for subjects on their cholesterol levels, body weight and other metabolic parameters, as well as a potential augmentation of the anti-psychotic effect of olanzapine.

This is a multi-centre randomised, double-blind, placebo-controlled, parallel-group pilot study. There will be two groups of subjects (GWP42003 plus GWP42004 (40:1 ratio) and placebo), with a treatment duration of 6 weeks as well as a baseline period of variable length and one week follow-up. The two treatment groups will be randomised equally.

In order to be eligible for enrollment in this study, subjects will need to be aged 18 years and above and be clinically diagnosed with functional psychosis and receiving olanzapine treatment for no more than 3 months with evidence of weight gain attributable to olanzapine treatment.

Eligible subjects will enter the study at a screening visit (Visit 1) and commence a baseline period. Subjects will also be assessed at Visit 2 for further weight gain during the baseline period. The baseline period is flexible in length to allow time for this weight gain to be achieved and also for the olanzapine dose to be stabilised. If eligible the subject will be randomised into the 6-week treatment phase. There are a total of 6 visits in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis (DSM-IV) of schizophrenia or functional psychosis including schizophreniform and acute psychosis with schizophrenia symptoms
* Receiving olanzapine treatment for no more than 3 months
* The dose of olanzapine is stable for at least 2 weeks prior to randomisation (Visit 2) and subject is willing to maintain a stable dose of olanzapine for the duration of the study
* Evidence of weight gain in the last 3 months attributable to olanzapine, prior to screening (Visit 1). Wherever possible, investigator must exclude other possible causes of weight gain, such as change in exercise, diet, or other illnesses
* Each subject must have further weight gain attributable to olanzapine, in the baseline period (between Visits 1 and 2) no more than 5 months subsequent to commencement of olanzapine treatment
* Willing to maintain a stable dose of any concomitant medications, and have been on a stable dose for a minimum of 6 weeks (with the exception of olanzapine)
* No changes in diet or exercise for 6 weeks prior to screening (Visit 1) and subject agrees to maintain stability, for the duration of the study (in the opinion of the investigator)

Exclusion Criteria:

* Subject has Axis I (DSM-IV) diagnosis of schizoaffective disorder;
* Subject has drug induced or toxic psychosis (in the opinion of the investigator)
* Subject presents with a clinical picture and/ or history that is consistent with delirium, dementia, amnesia or other cognitive disorder; bipolar disorder or major depression
* Subject has a significant history of anxiety, suicidal ideation or self-harm based on history or routine psychiatric status examination (in the opinion of the investigator)
* Subject has an unstable thyroid pathology (including hypo or hyperthyroidism), within the past six months (in the opinion of the investigator)
* Subject has a history of neuroleptic malignant syndrome;
* Subject requires or has had electroconvulsive therapy (ECT) treatment in the 2 month period prior to randomisation (Visit 2)
* Subject has a clinical diagnosis of diabetes
* Subject is taking insulin (i.e. they are insulin dependent) or have had insulin within 6 months prior to the screening visit (Visit 1);
* Any known or suspected history of (in the opinion of the investigator):
* alcohol or substance abuse
* epilepsy or recurrent seizures
* Any known or suspected history of depression sufficient to require treatment or disrupt ordinary life (excluding episodes of reactive depression - in the opinion of the investigator)
* BDI Score ≥ 15 (at Visit 1 or 2)
* Clinically significant cardiac, renal or hepatic impairment in the opinion of the investigator
* Genetic dyslipidaemic condition in the opinion of the investigator
* Female patients of child-bearing potential and male patients whose partner is of child-bearing potential, unless willing to ensure that they or their partner use effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (however, a male condom should not be used in conjunction with a female condom as this may not prove effective)
* Travel outside the country of residence planned during the study treatment period
* Having received olanzapine treatment continuously for more than 3 months prior to screening (Visit 1)
* Received an Investigational Medicinal Product within the 90 days before the screening visit (Visit 1)
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, influence the result of the study, or the subject's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PI, Principal Investigator — South London; PI, Principal Investigator — Birmingham; PI, Principal Investigator — West London; PI, Principal Investigator — Leicester; PI, Principal Investigator — Surrey; CI, Principal Investigator — Oxford
Locations (6):
- United Kingdom (6):
  - Birmingham
  - Leicester
  - Oxford
  - South London
  - Surrey
  - West London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was problematic due to the restrictive entry criteria (one subject screened in the first 5 months). Even after implementation of a protocol amendment to improve recruitment, only 12 subjects were screened and two randomised. It was decided that it would be impossible to complete the study in a meaningful timeframe so it was terminated.
Pre-assignment Details: There were a high proportion of screen failures due to most subjects failing to comply with one or more of the eligibility criteria.
Groups:
- GWP42003 : GWP42004 (40:1): Active study medication as 4 capsules GWP42003 and 2 capsules GWP42004 once daily.
- Placebo: Taken as 6 capsules, matched to taste and look like the active study medication.
Period: Overall Study
Arm/Group | GWP42003 : GWP42004 (40:1) | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only two subjects of a planned 60 were randomised due to early termination of the study due to problems with recruitment.
Groups:
- Placebo: Taken as 6 capsules once daily, matched to taste and look like the active study medication.
- Total: Total of all reporting groups
Arm/Group | GWP42003 : GWP42004 (40:1) | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (NA) — Only 1 participant contributed to the mean. | 37 (NA) — Only 1 participant contributed to the mean. | 30.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Bodyweight.
Description: Efficacy of a 40:1 ratio of GWP42003:GWP42004 compared with placebo in the change from baseline in body weight after 42 days (6 weeks) in subjects currently being treated with olanzapine for schizophrenia or other non-affective psychosis.
Time Frame: 6 weeks from Baseline.
Measure: Number; unit: Kg
Arm/Group | GWP42003 : GWP42004 (40:1) | Placebo
Number analyzed (Participants) | 1 | 1
Kg | 3.6 | 1

ADVERSE EVENTS:
Arm/Group | GWP42003 : GWP42004 (40:1) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GWP42003 : GWP42004 (40:1) (N=1) | Placebo (N=1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) — AEs assessed and noted a each study visit.

LIMITATIONS AND CAVEATS:
Early termination due to low subject recruitment meant only two subjects were randomised; one to active and the other to placebo. Only safety data of these two subjects has been reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be submitted to GW for corporate review before release. The principal investigators must then incorporate all reasonable comments made by GW into the publication.

GW also reserve the right to delay the submission of such information by up to six months from the date of first submission to them in order to allow them to take steps to protect proprietary information where applicable.